CLINICAL TRIAL: NCT03654586
Title: A Randomized-controlled Experiment on the Effects of Sugary Drink Warning Labels
Brief Title: Effects of Sugary Drink Warning Labels
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely during COVID-19 outbreak
Sponsor: University of Pennsylvania (Other)
Collaborators: Drexel University (Other); New York University (Other); University of Connecticut (Other)
Responsible Party: Principal Investigator, Christina Roberto, PHD, Assistant Professor of Medical Ethics and Health Policy, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1R01DK111558-01A1 (NIH)
Record Dates: First submitted 2018-08-07; First posted 2018-08-31 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Diabetes; Weight Gain
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Weight Gain

STUDY DESIGN:
Intervention Model Description: There was no answer option for our study design, but factorial is most similar. Participants will be randomly assigned to one of four conditions described below.
  1. Calorie label (control) will display a "Calories per Bottle" label on all beverages, not just sugary drinks. This is modeled after the American Beverage Association's current "Clear on Calories" labels.
  2. Text warning labels will display the following text on sugary beverages: WARNING: drinking beverages with added sugars contributes to obesity, diabetes, and tooth decay
  3. Sugar graphic warning labels will display the same text as "text warning labels" along with graphics depicting the amount of sugar in the beverage
  4. Health graphic warning label will display the same text as "text warning labels" along with graphics depicting the potential negative health consequences of over-consuming sugary drinks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Calorie label (Active Comparator): Calorie label (control) will display a "Calories per Bottle" label on all beverages, not just sugary drinks. This is modeled after the American Beverage Association's current "Clear on Calories" labels.
  Interventions: Behavioral: Sugary drink warning labels
- Text warning label (Experimental): Text warning labels will display the following text on sugary beverages: WARNING: drinking beverages with added sugars contributes to obesity, diabetes, and tooth decay
  Interventions: Behavioral: Sugary drink warning labels
- Sugar graphic warning label (Experimental): Sugar graphic warning labels will display the same text as "text warning labels" along with graphics depicting the amount of sugar in the beverage
  Interventions: Behavioral: Sugary drink warning labels
- Health graphic warning label (Experimental): Health graphic warning label will display the same text as "text warning labels" along with graphics depicting the potential negative health consequences of over-consuming sugary drinks.
  Interventions: Behavioral: Sugary drink warning labels

INTERVENTIONS:
Behavioral: Sugary drink warning labels — The description of each intervention appears in the descriptions of the experimental arms.

SUMMARY:
The primary objective of this study is to determine to what degree sugary drink warning labels increase consumers' knowledge about the potential health harms of sugary drinks and reduce sugary drink intake. The study is designed to answer three additional questions: 1) Do some warning labels work better than others? 2) What is the effect of warning labels over time? 3) If warning labels influence behavior, is it because they increase knowledge or simply provide a salient reminder that some drinks are less healthy? This study will test the effect of repeated exposure to warning labels on total calories purchased over time and assess whether knowledge or salience better explain label effects.

ELIGIBILITY:
Inclusion Criteria: Participants must:

* be a primary caregiver of a child under 12 years old;
* be ≥18 years old;
* read and speak English;
* drink sugary drinks at least twelve times per month (~three times per week) and have a child who does the same
* be the primary grocery shopper for their family;
* have regular internet access.

Exclusion Criteria:

* not a primary caregiver of a child under 12 years old
* <18 years old
* cannot read and speak English
* does not drink sugary drinks at least 12 times per month and have a child who does the same
* is not the primary grocery shopper for their family
* does not have regular internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Total calories purchased | four weeks
  total calories purchased over four weeks in an online store.
Total calories purchased in last two weeks of study | six weeks
  total calories purchased in the last two weeks of the study, after the labels are removed from the store.

SECONDARY OUTCOMES:
Noticing the calorie label | These will be assessed at one time point at the end of the 6-week study
  We will compare the percentage reporting "yes," "no," or "I don't know" to the question: "When you were buying beverages in the online store, did you notice any calorie labels next to the beverages?"
Perceived calorie label influence | These will be assessed at one time point at the end of the 6-week study
  We will compare the percent responding "yes", "no," or "I did not notice any labels" in response to the question of whether the calorie label influenced their purchase.
Noticing the warning label | These will be assessed at one time point at the end of the 6-week study
  We will compare the percent responding "yes", "no," or "I did not notice any labels" in response to the question, "When you were buying beverages in the online store, did you notice any warning labels next to the beverages?"
Perceived warning label influence | These will be assessed at one time point at the end of the 6-week study
  We will compare the percent responding "yes", "no," or "I did not notice any labels" in response to the question of whether the warning label influenced their purchase.
Label message recall | These will be assessed at one time point at the end of the 6-week study
  Participants will be prompted to remember the message on the warning labels in response to the following question: "If you saw warning labels, please type what you think the label said in the text box below." If participants cannot remember what the label said, they will be encouraged to respond with their best guess. If participants believe they did not see a label, they will be instructed to respond with "I did not see a warning label." We will examine the percent correctly recalling the label message.
Likelihood of buying the beverage | These will be assessed at one time point at the end of the 6-week study
  Item: "How likely are you to buy this beverage in the next 4 weeks?" Responses will be measured on a 5-point Likert scale ranging from 'Not at all' to 'Extremely'.
Parent affect around serving non-sugary beverages | These will be assessed at one time point at the end of the 6-week study
  This scale measures parents' affect toward serving their child non-sugary beverages. We will create this outcome by averaging responses to the following two questions separately for all non-sugary beverages: "Serving this beverage to my child would make me feel like a good parent" AND "Serving this beverage to my child would make me feel like I am doing something good for my child." These will be measured on 5-point Likert scales. The average non-sugary response for each participant will yield a scale ranging 1 (worse outcome) to 5 (better outcome).
Parent affect around serving sugary beverages | These will be assessed at one time point at the end of the 6-week study
  This scale measures parents' affect toward serving their child sugary beverages. We will create this outcome by averaging responses to the following two questions separately for all sugary beverages: "Serving this beverage to my child would make me feel like a good parent" AND "Serving this beverage to my child would make me feel like I am doing something good for my child." These will be measured on 5-point Likert scales. The average sugary response for each participant will yield a scale ranging 1 (better outcome) to 5 (worse outcome).
Enjoyment of non-sugary beverages | These will be assessed at one time point at the end of the 6-week study
  This scale measures parents' enjoyment of non-sugary beverages. We will create this outcome by averaging responses to "How delicious is this beverage?" separately for all non-sugary beverages. These will be measured on 5-point Likert scales. The average non-sugary response for each participant will yield a scale ranging 1 (worse outcome) to 5 (better outcome).
Enjoyment of sugary beverages | These will be assessed at one time point at the end of the 6-week study
  This scale measures parents' enjoyment of sugary beverages. We will create this outcome by averaging responses to "How delicious is this beverage?" separately for all sugary beverages. These will be measured on 5-point Likert scales. The average sugary response for each participant will yield a scale ranging 1 (better outcome) to 5 (worse outcome).
Healthiness of non-sugary beverages | These will be assessed at one time point at the end of the 6-week study
  This scale measures parents' belief in the healthiness of non-sugary beverages. We will create this outcome by averaging responses to "How healthy is this beverage?" separately for all non-sugary beverages. These will be measured on 5-point Likert scales. The average non-sugary response for each participant will yield a scale ranging 1 (worse outcome) to 5 (better outcome).
Healthiness of sugary beverages | These will be assessed at one time point at the end of the 6-week study
  This scale measures parents' belief in the healthiness of sugary beverages. We will create this outcome by averaging responses to "How healthy is this beverage?" separately for all sugary beverages. These will be measured on 5-point Likert scales. The average sugary response for each participant will yield a scale ranging 1 (better outcome) to 5 (worse outcome).
Non-sugary beverage influence on child's energy and focus | These will be assessed at one time point at the end of the 6-week study
  This scale measures parents' belief that drinking non-sugary beverages improves their child's energy and focus. We will create this outcome by averaging responses to the following two questions separately for all non-sugary beverages: "Drinking this beverage often would make my child feel energized" and "Drinking this product often would help my child focus at school." These will be measured on 5-point Likert scales. The average non-sugary response for each participant will yield a scale ranging 1 (worse outcome) to 5 (better outcome).
Sugary beverage influence on child's energy and focus | These will be assessed at one time point at the end of the 6-week study
  This scale measures parents' belief that drinking sugary beverages improves their child's energy and focus. We will create this outcome by averaging responses to the following two questions separately for all sugary beverages: "Drinking this beverage often would make my child feel energized" and "Drinking this product often would help my child focus at school." These will be measured on 5-point Likert scales. The average sugary response for each participant will yield a scale ranging 1 (better outcome) to 5 (worse outcome).
Non-sugary drink health beliefs and risk perceptions index | These will be assessed at one time point at the end of the 6-week study
  This scale measures parents' health beliefs and risk perceptions about their child's drinking non-sugary beverages. We will create this outcome by averaging the responses to the following health perception questions prompted with the statement "If my child drank this beverage often it would…" across all non-sugary beverages. The statements end with the following health belief and risk perception language: "cause my child to gain weight," "increase my child's risk of heart disease," "increase my child's risk of diabetes," "increase my child's risk of cancer," and "help my child live a healthier life." Responses to questions about weight gain, heart disease, diabetes, and cancer will be reverse coded, so higher scores on the index will indicate a stronger positive health perception of the non-sugary beverages. All variables will be measured on a 5-point Likert scale. The average non-sugary response for each participant will yield a scale ranging 1 (worse outcome) to 5 (better outcome).
Sugary drink health beliefs and risk perceptions index | These will be assessed at one time point at the end of the 6-week study
  This scale measures parents' health beliefs and risk perceptions about their child's drinking sugary beverages. We will create this outcome by averaging the responses to the following health perception questions prompted with the statement "If my child drank this beverage often it would…" across all sugary beverages. The statements end with the following health belief and risk perception language: "cause my child to gain weight," "increase my child's risk of heart disease," "increase my child's risk of diabetes," "increase my child's risk of cancer," and "help my child live a healthier life." Responses to questions about weight gain, heart disease, diabetes, and cancer will be reverse coded, so higher scores on the index will indicate a stronger positive health perception of the sugary beverages. All variables will be measured on a 5-point Likert scale. The average sugary response for each participant will yield a scale ranging 1 (better outcome) to 5 (worse outcome).
Estimate of calories per non-sugary drink bottle | These will be assessed at one time point at the end of the 6-week study
  This variable will be the average across all responses to non-sugary beverages measured continuously based on open-ended text box provided to participants. Responses will be limited to a maximum of 4-digits. Numbers closer to the true average will be the better outcome.
Estimate of calories per sugary drink bottle | These will be assessed at one time point at the end of the 6-week study
  This variable will be the average across all responses to sugary beverages measured continuously based on open-ended text box provided to participants. Responses will be limited to a maximum of 4-digits. Numbers closer to the true average will be the better outcome.
Estimate of teaspoons of added sugar per non-sugary drink bottle | These will be assessed at one time point at the end of the 6-week study
  This variable will be an average across all non-sugary beverages of a 4-point Likert scale ranging from 'None' (1; better outcome) to 'A lot' (4; worse outcome).
Estimate of teaspoons of added sugar per sugary drink bottle | These will be assessed at one time point at the end of the 6-week study
  This variable will be an average across all sugary beverages of a 4-point Likert scale ranging from 'None' (1; worse outcome) to 'A lot' (4; better outcome).
Perceived amount of sugar | These will be assessed at one time point at the end of the 6-week study
  Item: "Do you think this amount of sugar for your child is…?" This variable will be measured on a 3-point Likert scale ranging from "too little" (1; worse outcome) to "too much" (3; better outcome)
Label trust | These will be assessed at one time point at the end of the 6-week study
  Item: "How much do you trust the information on this label?". Responses will be measured on a 5-point Likert scale.
Label purchase influence | These will be assessed at one time point at the end of the 6-week study
  Item: "When you saw this label next to an item in the store, to what extent were you less or more likely to buy the item?" The responses will be measured on a 5-point Likert scale.
Positive and negative reactions to the label | These will be assessed at one time point at the end of the 6-week study
  We will compare the percentage of people that had a predominantly positive reaction to the label (percentage of people that said the warning label predominantly made them feel hopeful or happy. We will average across these ratings and define this as an average score >3 on a 1-5 Likert scale)
Negative reactions to the label | These will be assessed at one time point at the end of the 6-week study
  We will compare the percentage of people that had a predominantly negative reaction to the label (percentage of people that said the warning label predominantly made them feel depressed, fearful, guilty, discouraged, annoyed, scared, disgusted or grossed out, sad, angry, or afraid. We will average across these ratings and define this as an average score >3 on a 1-5 Likert scale)
Newest vital sign measure | These will be assessed at one time point at the end of the 6-week study
  Participants will be shown a nutrition label and asked to answer some questions that will require them to read and understand the information presented on the label. This is a publically available, validated assessment. We will examine this as a moderator of label effects.

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Roberto, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Blockley Hall, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share a de-identified dataset via an online data storage website (e.g., open science framework, dataverse, research box)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be made available soon after the paper is published in a peer-reviewed journal.
Access Criteria: All researchers will be able to access the data